CLINICAL TRIAL: NCT05047471
Title: Healthy China - The Improvement Projects for the Screening Ability of Diabetes and Its Complications And for the Standardized Ability of Diagnosis and Treatment for Patients With Early Diabetic Nephropathy
Brief Title: To Improve the Ability of Early Screening and Diagnosis in Patients With Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yiming Mu (Other)
Responsible Party: Sponsor-Investigator, Yiming Mu, Director of department, Beijing Great Physician Commonweal Foundation
Organization: Beijing Great Physician Commonweal Foundation (Other)
Other Study IDs: 2021BY01
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Kidney Disease
Keywords: SGLT2 inhibitors; Diabetic Kidney Disease; Albuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a large-scale, multi-center, observational study. It is planned to establish a large database of 10,000 patients with type 2 diabetes mellitus to investigate the prevalence, awareness and screening rates of diabetes kidney disease (DKD), and provide real-world data on the efficacy and safety of sodium glucose cotransporter 2 inhibitors (SGLT2i) in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Among the various complications of diabetes mellitus, DKD is considered as a major threat and is one of the manifestations of diabetic microangiopathy. it is one of the main causes of death for patients with T2DM.

Albuminuria is the earliest manifestation of DKD, which is mostly asymptomatic at the early stage, if the albuminuria is poorly controlled, it may develop into clinical DKD. Therefore, it is very important to improve the patients' awareness of DKD, regularly screen early kidney diseases and use drugs rationally.

In order to promote the standardization of diagnosis and treatment of patients with DKD, improve the knowledge and screening rate of patients with DKD, help the formation of health literacy, healthy behavior and lifestyle, the investigators planned the study.

STUDY OBJECTIVES:

1. To understand the epidemiological disease burden of DKD in China, and to investigate the prevalence rate, awareness rate and screening rate of DKD;
2. To understand the treatment status of patients with DKD in China;
3. To provide real-world data on the efficacy and safety of SGLT2i in the treatment of DKD in China;

ELIGIBILITY:
Inclusion Criteria:

* It is known that patients with T2DM has a history of more than 12 months (the WHO1999 Standard) and is treated with at least one anti-diabetic agent.
* Gender and age: men and women who are at least 18 years old with informed consent.
* Patients are willing and able to provide written informed consent before participating in this study.

Exclusion Criteria:

* Type 1 diabetes mellitus (DM)
* Patients with severe ketosis, diabetic coma, severe infection or severe trauma
* Perioperative patients
* Patients with severe renal impairment and advanced nephropathy (eGFR < 45 ml/min/1.73m2)
* Renal transplant patients
* Patients are participating in or have participated in any other clinical trials in the past 3 months
* Any disease with a life expectancy of less than 2 years according to the clinical judgment of the investigator
* Pregnant or lactating women
* Patients judged by the investigator to be unsuitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous screening of type 2 diabetic patients from the endocrinology outpatients of 50 hospitals across the country
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of DKD | at the time of screening
  Prevalence of DKD (UACR > 30 mg/g); The prevalence of microalbuminuria (30 mg/g ≤ UACR ≤ 300 mg/g); The prevalence of massive proteinuria (UACR > 300 mg/g).
Awareness rate | at the time of screening
  Awareness rate=(The number of people who know their abnormal albuminuria)/(The number of people with diabetes mellitus complicated with albuminuria)
Screening rate | at the time of screening
  Screening rate=(The number of people @who have checked urine protein within one year)/(The number of people involved in total diabetes)
Prescription proportion of various anti-diabetic drugs for patients with DKD | at the time of screening
  Prescription ratio of a certain hypoglycemic agent =(The number of people using a certain hypoglycemic agent)/(Total number of DKD)
risk factors of albuminuria: medication categories | at the time of screening
  Assess whether taking different categories of medications is a risk factor for albuminuria
risk factors of albuminuria: Course of disease | at the time of screening
  It is defined as the years of diagnosis of diabetes. According to the "Date of Diagnosis" in the questionnaire collected during the screening, the course years of diabetes patients are divided into quartiles for evaluation
risk factors of albuminuria: Age | at the time of screening
  According to the "date of birth" in the questionnaire collected during the screening, the age of diabetic patients is divided into quartiles for evaluation
risk factors of albuminuria: Current smoking | at the time of screening
  According to the "Current smoking" in the questionnaire collected during the screening to evaluate whether smoking is the risk of albuminuria
risk factors of albuminuria: gender | at the time of screening
  According to the "gender" in the questionnaire collected during the screening to evaluate whether gender is the risk of albuminuria
risk factors of albuminuria: Drinking | at the time of screening
  According to the " Drinking " in the questionnaire collected during the screening to evaluate whether Drinking is the risk of albuminuria
risk factors of albuminuria: Glycosylated hemoglobin | at baseline
  Baseline glycosylated hemoglobin is divided into quartiles for evaluation
risk factors of albuminuria: Hypertension | at baseline
  It is defined as the adults' systolic blood pressure which is greater than or equal to 140mmHg and/or diastolic blood pressure which is greater than or equal to 90mmHg. "hypertension" and "non-hypertension" for evaluation
risk factors of albuminuria: Increase in Low density lipoprotein cholesterol (LDL-C) | at baseline
  It is defined as more than 3.37mmol/L, "elevated" and "normal" for evaluation

SECONDARY OUTCOMES:
MD of the change of UACR | at 6 months
  the mean difference of the change of UACR from baseline between SGLT2i and non-SGLT2i group
OR of the incidence of the adverse events | at 6 months
  the odds ratio of the incidence of the adverse events of interest during the 6-month observation period between SGLT2i and non-SGLT2i group

OTHER OUTCOMES:
MD of the Percentage change of HbA1c | at 6 months
  the mean difference of the Percentage change from baseline of HbA1c between SGLT2i group and non-SGLT2i group
MD the Percentage change from baseline of other laboratory test parameters of interest | at 6 months
  the mean difference of the Percentage change from baseline of other laboratory test parameters of interest in SGLT2i group and non-SGLT2i group

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mu, MD, Principal Investigator — The First Medical Center of Chinese PLA General Hospital
Locations (50):
- China (50):
  - Airport Area of Peking University Third Hospital, Beijing
  - Beijing Haidian Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital Yanqing Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Strategic Support Force Specialty Medical Center, Beijing
  - The 3th Medical Center of Chinese PLA General Hospital, Beijing
  - The 4th Medical Center of Chinese PLA General Hospital, Beijing
  - The 5th Medical Center of Chinese PLA General Hospital, Beijing
  - The 6th Medical Center of Chinese PLA General Hospital, Beijing
  - The 7th Medical Center of Chinese PLA General Hospital, Beijing
  - The 8th Medical Center of Chinese PLA General Hospital, Beijing
  - The First Medical Center of Chinese PLA General Hospital, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Guangzhou Red Cross Hospital, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Guiyang First People's Hospital, Guiyang
  - Guiyang Second People's Hospital, Guiyang
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital of Guizhou Medical University, Guiyang
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - NanjingNanjing Drum Tower Hospital( the Affiliated Hospital of Nanjing University Medical School), Nanjin
  - Nanjing First Hospital, Nanjing
  - Nantong First People's Hospital, Nantong
  - Qingdao Eighth People's Hospital, Qingdao
  - Qingdao Third People's Hospital, Qingdao
  - The Affiliated Hospital of Qingdao University, Qingdao
  - People's Hospital of Rizhao, Rizhao
  - Qingpu Branch of Zhongshan Hospital affiliated to Fudan University, Shanghai
  - Shanghai Minhang District Central Hospital, Shanghai
  - Shanghai Xuhui District Central Hospital, Shanghai
  - Wusong Hospital, Zhongshan Hospital affiliated to Fudan University, Shanghai
  - Zhongshan Hospital affiliated to Fudan University, Shanghai
  - Second Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Taizhou Second People's Hospita, Taizhou
  - Weihai Municipal Hospital, Weihai
  - Renmin Hospital of Wuhan University, Wuhan
  - The Central Hospital of Wuhan, Wuhan
  - Tongji Hospital, Tongji Medical College Of HUST, Wuhan
  - Wuhan No. 1 Hospital, Wuhan
  - Wuhan No. 3 Hospital, Wuhan
  - Wuhan No. 4 Hospital, Wuhan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Yixing People's Hospital, Yixing
  - Zhenjiang First People's Hospital, Zhenjiang
  - The Affiliated Hospital of Zunyi Medical University, Zunyi
  - Zunyi First People's Hospital, Zunyi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant level data and measurements including tables, figures, and appendices or supplementary material that support the results presented in a manuscript will be shared 6 months after publication.
Time Frame: starting 6 months after publication
Access Criteria: Researches should send a proposal to muyiming@301hospital.com.cn. If the proposal is methodologically sound, feasible and approved by the principal investigator, data requestor could gain access after signing a data access agreement.
URL: http://www.bgpcf.net

REFERENCES:
- [Background] Wen CP, Chang CH, Tsai MK, Lee JH, Lu PJ, Tsai SP, Wen C, Chen CH, Kao CW, Tsao CK, Wu X. Diabetes with early kidney involvement may shorten life expectancy by 16 years. Kidney Int. 2017 Aug;92(2):388-396. doi: 10.1016/j.kint.2017.01.030. Epub 2017 Jun 1. PMID 28577854
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] Cannon CP, Pratley R, Dagogo-Jack S, Mancuso J, Huyck S, Masiukiewicz U, Charbonnel B, Frederich R, Gallo S, Cosentino F, Shih WJ, Gantz I, Terra SG, Cherney DZI, McGuire DK; VERTIS CV Investigators. Cardiovascular Outcomes with Ertugliflozin in Type 2 Diabetes. N Engl J Med. 2020 Oct 8;383(15):1425-1435. doi: 10.1056/NEJMoa2004967. Epub 2020 Sep 23. PMID 32966714
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Bailey CJ, Gross JL, Hennicken D, Iqbal N, Mansfield TA, List JF. Dapagliflozin add-on to metformin in type 2 diabetes inadequately controlled with metformin: a randomized, double-blind, placebo-controlled 102-week trial. BMC Med. 2013 Feb 20;11:43. doi: 10.1186/1741-7015-11-43. PMID 23425012
- [Background] Strojek K, Yoon KH, Hruba V, Elze M, Langkilde AM, Parikh S. Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with glimepiride: a randomized, 24-week, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2011 Oct;13(10):928-38. doi: 10.1111/j.1463-1326.2011.01434.x. PMID 21672123
- [Background] Guo K, Zhang L, Zhao F, Lu J, Pan P, Yu H, Bao Y, Chen H, Jia W. Prevalence of chronic kidney disease and associated factors in Chinese individuals with type 2 diabetes: Cross-sectional study. J Diabetes Complications. 2016 Jul;30(5):803-10. doi: 10.1016/j.jdiacomp.2016.03.020. Epub 2016 Mar 17. PMID 27068269
- [Background] Shikata K, Kodera R, Utsunomiya K, Koya D, Nishimura R, Miyamoto S, Tajima N; JDCP study group. Prevalence of albuminuria and renal dysfunction, and related clinical factors in Japanese patients with diabetes: The Japan Diabetes Complication and its Prevention prospective study 5. J Diabetes Investig. 2020 Mar;11(2):325-332. doi: 10.1111/jdi.13116. Epub 2019 Sep 25. PMID 31317670
- [Background] Mok KY, Chan PF, Lai LKP, Chow KL, Chao DVK. Prevalence of diabetic nephropathy among Chinese patients with type 2 diabetes mellitus and different categories of their estimated glomerular filtration rate based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation in primary care in Hong Kong: a cross-sectional study. J Diabetes Metab Disord. 2019 Nov 15;18(2):281-288. doi: 10.1007/s40200-018-00382-y. eCollection 2019 Dec. PMID 31890652
- [Background] Jitraknatee J, Ruengorn C, Nochaiwong S. Prevalence and Risk Factors of Chronic Kidney Disease among Type 2 Diabetes Patients: A Cross-Sectional Study in Primary Care Practice. Sci Rep. 2020 Apr 10;10(1):6205. doi: 10.1038/s41598-020-63443-4. PMID 32277150
- [Background] Pollock C, Stefansson B, Reyner D, Rossing P, Sjostrom CD, Wheeler DC, Langkilde AM, Heerspink HJL. Albuminuria-lowering effect of dapagliflozin alone and in combination with saxagliptin and effect of dapagliflozin and saxagliptin on glycaemic control in patients with type 2 diabetes and chronic kidney disease (DELIGHT): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 Jun;7(6):429-441. doi: 10.1016/S2213-8587(19)30086-5. Epub 2019 Apr 13. PMID 30992195
- [Derived] Shi L, Xue Y, Yu X, Wang Y, Hong T, Li X, Ma J, Zhu D, Mu Y. Prevalence and Risk Factors of Chronic Kidney Disease in Patients With Type 2 Diabetes in China: Cross-Sectional Study. JMIR Public Health Surveill. 2024 Aug 30;10:e54429. doi: 10.2196/54429. PMID 39213031
- See also: Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition) — http://med.wanfangdata.com.cn/Paper/Detail?dbid=WF_QK&id=PeriodicalPaper_zhtnb202104005